CLINICAL TRIAL: NCT01565434
Title: Erythrocyte Complement Receptor 1 and Alzheimer Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Purpose: Screening
Other Study IDs: PA11014
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2012-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: CR1 impact

SUMMARY:
Main objective: investigate whether a functional polymorphism of CR1 (length, number of binding sites in C4b C3b, erythrocyte density, rate of soluble CR1 ...) so determined genetic or acquired, is a susceptibility factor for the disease Alzheimer's.

ELIGIBILITY:
Inclusion Criteria:

* caucasians people with a Alzheimer dementia defined on DSMIV criteria for patients and without Alzheimer disease for control subjects

Exclusion Criteria:

* diseases modifying CR1 physiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-02; Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de REIMS, Reims, France

REFERENCES:
- [Background] Mahmoudi R, Kisserli A, Novella JL, Donvito B, Drame M, Reveil B, Duret V, Jolly D, Pham BN, Cohen JH. Alzheimer's disease is associated with low density of the long CR1 isoform. Neurobiol Aging. 2015 Apr;36(4):1766.e5-1766.e12. doi: 10.1016/j.neurobiolaging.2015.01.006. Epub 2015 Jan 9. PMID 25666996
- [Result] Mahmoudi R, Feldman S, Kisserli A, Duret V, Tabary T, Bertholon LA, Badr S, Nonnonhou V, Cesar A, Neuraz A, Novella JL, Cohen JHM. Inherited and Acquired Decrease in Complement Receptor 1 (CR1) Density on Red Blood Cells Associated with High Levels of Soluble CR1 in Alzheimer's Disease. Int J Mol Sci. 2018 Jul 25;19(8):2175. doi: 10.3390/ijms19082175. PMID 30044434